CLINICAL TRIAL: NCT07195474
Title: Effect of Daily Yogurt Smoothies on Neurocognitive Function in Children
Brief Title: Smoothie Program for Achieving and Resilient Kids
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Professor in Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00027677
Record Dates: First submitted 2025-08-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Executive Functions (EF); Microbiome; Dietary Quality
Keywords: Cognitive Function; daily yogurt smoothies intake; gut and brain health; hippocampal-dependent memory; dose-dependent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, Research Assistants (RAs) responsible for administering tasks and collecting data (e.g., behavioral assessments, fNIRS recordings) are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 daily yogurt smoothie (Experimental): Children will have the experimental doses of yogurt smoothies (1x daily) for 4 weeks. (93 mL and ~70 kcal)
  Interventions: Dietary Supplement: Yogurt Smoothie (1 per day)
- 2 daily yogurt smoothies (Experimental): Children will have the experimental doses of yogurt smoothies (2x daily) for 4 weeks. (186 mL and ~140 kcal)
  Interventions: Dietary Supplement: Yogurt Smoothie (2 per day)
- daily fruit juice control (Active Comparator): Children will have the fruit juice control (1 juice per day) for 4 weeks. (isocaloric fruit juice ~140 kcal)
  Interventions: Dietary Supplement: Fruit Juice Control

INTERVENTIONS:
Dietary Supplement: Yogurt Smoothie (1 per day) — Children consume one yogurt smoothie per day for 4 weeks (93 mL and ~70 kcal).
  Arms: 1 daily yogurt smoothie
Dietary Supplement: Yogurt Smoothie (2 per day) — Children consume two yogurt smoothies per day for 4 weeks (186 mL and ~140 kcal).
  Arms: 2 daily yogurt smoothies
Dietary Supplement: Fruit Juice Control — Children consume one fruit juice per day for 4 weeks (~140 kcal, isocaloric with 2 yogurt smoothie).
  Arms: daily fruit juice control

SUMMARY:
The proposed study will examine whether eating yogurt every day can improve brain and gut health in children. Prior research suggests that yogurt may support cognitive functions like self-control, but more studies are needed to confirm this. The study will follow 60 children from Central Pennsylvania, ages 7 to 9, who will be randomly assigned to drink either fruit juice (control group) or yogurt smoothies once or twice a day for four weeks.

Researchers will compare how different amounts of yogurt affect children's thinking skills (like memory and focus), brain activity, and gut bacteria. These changes will be measured through brain scans, computer-based thinking tasks, surveys, and stool samples. The study will also collect information about children's overall diet. The goal is to find out if yogurt can support healthy brain and gut development and to determine the right amount to include in a child's daily diet. Results will help guide future research on how nutrition supports children's health.

DETAILED DESCRIPTION:
This study is a randomized, between group, dose-response study. Children will be randomly assigned to either receive the control (fruit juice) or a dosage of the experimental yogurt smoothie (1x versus 2x daily) for 4 weeks. Blinding will be established so that researchers do not know which group children are assigned to and families do not know which smoothie is expected to change outcomes. Children will be advised to minimize additional consumption of fermented dairy during the intervention (besides the yogurt provided).

Outcomes will be measured at 2 timepoints: immediately before and immediately following the exposure (2 laboratory visits). The visits will take place around 4 weeks apart. In each visit, child participants will undergo a series of tasks, including a Stop Signal Task (SST), a Flanker Task, the Wide Range Assessment of Memory and Learning (WRAML3), the Delis-Kaplan Executive Function System (D-KEFS), the Weschler Abbreviated Scale of Intelligence (WASI-II), and the N-back test. During the N-back test, participants will wear an fNIRS cap to measure and record localized brain activity. Skin carotenoid levels will also be measured using the Veggie Meter. Throughout each visit, the parent participant will complete a series of questionnaires that assess family demographics, home food security, child behavior and temperament, child executive function, family food behaviors, child pubertal development, and beverage consumption frequency. Between the two visits, along with the consumption of the juice or yogurt each day, child participants will complete a weekly food log survey. Parent participants will also complete weekly surveys that assess home food inventory, food and beverage consumption practices, and child behavior. Additionally, parent participants will be asked to collect a fecal sample from their child 1-2 nights before each visit with a provided fecal sample collection kit.

ELIGIBILITY:
Inclusion Criteria:

* Children should be of good health, without presence of any metabolic, gastrointestinal, or developmental disorders (e.g., ADHD, autism, etc.).
* Children should not be taking medications that impact appetite or cognitive function.
* Children must be willing to consume and report liking the fermented dairy smoothie.
* Children should be between the ages of 7-9 years-old at enrollment.
* Children should speak English fluently.

Exclusion Criteria:

* They are not within the age requirements (< 7 years-old or > 9 years-old) at baseline.
* They have known emotional or cognitive delays, so that we can be assured that they understand the procedures.
* They do not speak English fluently.
* They have parentally reported medical problems that affect the digestive system or ability to eat yogurt (e.g., lactose intolerance, food allergies, Crohn's disease, Celiac disease, Esophagitis) and/or are taking a prescription medication that may affect appetite (e.g., Ritalin, methylphenidate, Adderall XR, Concerta, Vyvanse, etc.).
* They are not from families of rural communities (assessed by National Center for Education Statistics local classifications).
* Their parent is unable to attend the study visits.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive and Brain Responses to Yogurt Smoothie Intake | Baseline and up to average of 4 weeks
  The investigators will use standardized cognitive tests and functional near-infrared spectroscopy (fNIRS) to assess the effects of nutritional beverages, on executive function and hippocampal-dependent memory in children.
Prefrontal Cortex Activation During Working Memory After Yogurt Smoothie Intake | Baseline and up to average of 4 weeks
  The investigators will use fNIRS to assess prefrontal cortex activation while children complete a working memory task, comparing the effects of nutritional beverages.
Gut Microbiome and Executive Function Responses | Baseline and up to average of 4 weeks
  Fecal samples will be collected at multiple time points to analyze changes in the gut microbiome composition and metabolome. These changes will be correlated with improvements in child executive function (EF) and prefrontal cortex (PFC) activation.
Prefrontal Cortex Activation During Working Memory After Yogurt Smoothie Intake | Baseline and up to average of 4 weeks
  Working memory will be measured using the WRAML3 (Wide Range Assessment of Memory and Learning, Third Edition).

SECONDARY OUTCOMES:
Child anthropometrics | Baseline and up to average of 4 weeks
  Height and weight will be measured every week using a stadiometer scale. From these, BMI (Body Mass Index) will be calculated and converted to BMI z-score and BMI-for-age and sex percentile
Amount of smoothies leftover | Baseline and up to average of 4 weeks
  The remaining smoothies will be collected and weighed (gram amount not consumed), and parents will complete a questionnaire to log consumption.
Change in Emotional Symptoms Score (SDQ) | Every week
  Weekly parent-completed Strengths and Difficulties Questionnaire (SDQ) reporting emotional symptoms subscale, assessing 25 positive and negative behaviors
Dietary intake and quality | Assessed weekly
  Dietary intake will be assessed using two 24-hour dietary recalls per week (one weekday and one weekend day), completed with parental assistance through the ASA24 (Automated Self-Administered 24-hour Dietary Assessment Tool).
Pubertal stage | Pre-exposure
  Child Tanner stage will be reported by parents at baseline using the Tanner Staging Questionnaire (male or female).
Measures of carotenoids | Baseline and up to average of 4 weeks
  The investigators will use a Veggie Meter. It's a device that non-invasively measures the amount of carotenoids in a person's skin, which serves as an indicator of their fruit and vegetable consumption.
Incidence of Gastrointestinal Adverse Events | Every day
  Parents will complete a daily survey reporting the presence or absence of gastrointestinal symptoms (constipation, diarrhea, abdominal pain, bloating, nausea). Each symptom will be recorded as present/absent, and frequency will be assessed.
Acceptability of the Intervention | Every day
  Parents will complete a daily survey rating the acceptability of the intervention. Acceptability will be assessed using a Likert scale (e.g., 1 = not acceptable, 5 = highly acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Metabolic Kitchen and Children's Eating Behavior Lab, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drucker H, Wolcott RB. Gingival tissue management with Class V restorations. J Am Acad Gold Foil Oper. 1970 Apr;13(1):34-8. No abstract available. PMID 5267299
- [Background] Steiger E. Home parenteral nutrition. Components, application, and complications. Postgrad Med. 1984 May;75(6):95-102. doi: 10.1080/00325481.1984.11716310. PMID 6425815
- [Background] Pearce AL, Mackey E, Cherry JBC, Olson A, You X, Magge SN, Mietus-Snyder M, Nadler EP, Vaidya CJ. Effect of Adolescent Bariatric Surgery on the Brain and Cognition: A Pilot Study. Obesity (Silver Spring). 2017 Nov;25(11):1852-1860. doi: 10.1002/oby.22013. PMID 29086502
- [Background] Cravener TL, Schlechter H, Loeb KL, Radnitz C, Schwartz M, Zucker N, Finkelstein S, Wang YC, Rolls BJ, Keller KL. Feeding Strategies Derived from Behavioral Economics and Psychology Can Increase Vegetable Intake in Children as Part of a Home-Based Intervention: Results of a Pilot Study. J Acad Nutr Diet. 2015 Nov;115(11):1798-807. doi: 10.1016/j.jand.2015.03.024. Epub 2015 May 23. PMID 26014476